CLINICAL TRIAL: NCT01820923
Title: Study on the Use of Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation to Promote Diagnosis, Prognosis and Innovative Rehabilitation in Patients in Vegetative and Minimally Conscious State.
Brief Title: Transcranial Brain Stimulation in Vegetative State Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Marianna Cavinato, PhD, IRCCS San Camillo, Venezia, Italy
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011.04; 288/08 (Other Grant/Funding Number: Regional research funding)
Record Dates: First submitted 2013-03-14; First posted 2013-03-29 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Vegetative State; Minimally Conscious State
MeSH Terms: conditions — Persistent Vegetative State | interventions — Transcranial Direct Current Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brain stimulation (Experimental): Brain stimulation will consist of 4 types of intervention:
  * real transcranial direct current stimulation (two weeks, five days a week)
  * a week of wash-out
  * Sham transcranial direct current stimulation (two weeks, five days a week)
  * two weeks of wash-out
  * real repetitive transcranial magnetic stimulation (two weeks, four days a week)
  * a week of wash-out
  * Sham repetitive transcranial magnetic stimulation (two weeks, three days a week)
  Stimulations will be counterbalanced between patients.
  Interventions: Device: Transcranial direct current stimulation (tDCS); Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Transcranial Direct Current Stimulation (SHAM); Device: Repetitive Transcranial Magnetic Stimulation (SHAM)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — 2 mA of intensity, 20 minutes of stimulation over the left fronto-temporal prefrontal cortex.
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Frequency of stimulation: 10Hz. Interstimulus interval: 1 min. Number of stimuli per session: 300. Number of sessions per week: 4 Total number of stimuli: 1.200
Device: Transcranial Direct Current Stimulation (SHAM) — The electrodes of stimulation will be applied in the left fronto-temporal prefrontal cortex, but the device will be turned off.
Device: Repetitive Transcranial Magnetic Stimulation (SHAM) — The coil will be applied on the left fronto-temporal prefrontal cortex, but the device will be turned off.

SUMMARY:
The aim of this study is to determine whether transcranial brain stimulations, such as repetitive transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS), are effective in terms of EEG coherence and clinical changes in patients in vegetative and minimally conscious state.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of vegetative state od minimally conscious state defined by the Disability Rating Scale with a score between 17 and 29.
* Age between 18 and 65 years.
* Time from the lesion: more than 4 months.
* Stable clinical condition.
* written consent fron the legal administrator of the patient.

Exclusion Criteria:

* Presence of epileptiform activity on EEG.
* Previous history of epilepsy.
* Extensive hemorrhage or ischemia.
* Metallic clips or intracranial implants.
* Pacemaker e Baclofen infusion.
* Presence of drugs influencing arousal or awareness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
EEG coherence analysis | Change from baseline EEG coherence at the end of brain stimulation (two weeks)
  EEG will be filtered between 0.5 and 30Hz by elliptic filters. Fast Fourier Transformation will be performed on 2 sec-epochs. For each stimulation site, coherence values will be estimated within four frequency bands: Delta (0.5-3.5 Hz), Theta (4-7.5 Hz), Alpha (8-12.5 Hz), and Beta (13-30 Hz). Each coherence map will be proportionally thresholded, preserving 50% of the strongest coherence values, to produce a weighted adjacency matrix. The estimated functional connectivity patterns will be characterized by means of two global network metrics derived from graph theory: modularity and global efficiency. Modularity measures how the network is organized into modules with high level clustering. Global efficiency measures how efficient the network is in exchanging information at the global level.

SECONDARY OUTCOMES:
Disability Rating Scale | Change from baseline DRS scale at the end of brain stimulation (two weeks)

OTHER OUTCOMES:
Western Neuro Sensory Stimulation Profile (WNSSP) | Change from baseline WNSSP scale at the end of brain stimulation (two weeks)
  This scale is developed to assess cognitive function in severely impaired head-injured adults and to monitor and predict change in slow-to-recover patients.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Piccione, MD, Study Director — San Camillo Foundation
Locations (1):
- IRCCS San Camillo Foundation, Venice, Venice, Italy

REFERENCES:
- [Background] Giacino J, Fins JJ, Machado A, Schiff ND. Central thalamic deep brain stimulation to promote recovery from chronic posttraumatic minimally conscious state: challenges and opportunities. Neuromodulation. 2012 Jul;15(4):339-49. doi: 10.1111/j.1525-1403.2012.00458.x. Epub 2012 May 24. PMID 22624587
- [Result] Piccione F, Cavinato M, Manganotti P, Formaggio E, Storti SF, Battistin L, Cagnin A, Tonin P, Dam M. Behavioral and neurophysiological effects of repetitive transcranial magnetic stimulation on the minimally conscious state: a case study. Neurorehabil Neural Repair. 2011 Jan;25(1):98-102. doi: 10.1177/1545968310369802. Epub 2010 Jul 20. PMID 20647501